CLINICAL TRIAL: NCT05344911
Title: Comparison of Postoperative Pain Application of Alfentanil or Remifentanil in TIVA Undergoing Functional Endoscopic Sinus Surgery
Brief Title: Comparison of Postoperative Pain Application of Alfentanil or Remifentanil in TIVA
Acronym: TIVA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: xijing2022-0410
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Pain
Keywords: functional endoscopic sinus surgery; postoperative pain; afentanil or remifentanil
MeSH Terms: conditions — Pain, Postoperative | interventions — Alfentanil; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- remifentanil (Active Comparator): Anesthesia maintenance：target-controlled infusion of propofol combined with remifentanil）
  Interventions: Drug: Propofol combined with remifentanil
- alfentanil (Experimental): Anesthesia maintenance：target-controlled infusion of propofol combined with afentanil
  Interventions: Drug: Propofol combined with alfentanil

INTERVENTIONS:
Drug: Propofol combined with alfentanil — Anesthesia induction: midazolam 0.02 mg/kg, propofol（TCI） 3 μ g/mL, alfentanil 20 μ g/kg and rocuronium 0.6 mg/kg . Anesthesia maintenance: target-controlled infusion of propofol combined with alfentanil(0.5-2ug/kg/min)
  Arms: alfentanil
Drug: Propofol combined with remifentanil — Anesthesia induction: midazolam 0.02 mg/kg, propofol（TCI） 3 μ g/mL, remifentanil 1μ g/kg and rocuronium 0.6 mg/kg . Anesthesia maintenance: target-controlled infusion of propofol combined with remifentanil(0.1-0.3ug/kg/min)
  Arms: remifentanil

SUMMARY:
Total intravenous anesthesia (TIVA) is maintained by intermittent or continuous combined intravenous injection of a variety of short-acting intravenous anesthetics, which can provide safe and rapid induction, maintenance and termination of general anesthesia. It has a slight effect on respiration and circulation, strong controllability, short anesthetic recovery time, reduced postoperative nausea and vomiting (PONV) and quick discharge time, so it has been widely used in clinic. Functional endoscopic sinus surgery is a common method for the treatment of sinusitis and other diseases. The trauma of this operation is less. The use of TIVA during the operation can reduce the bleeding in the surgical field and is beneficial to the recovery of patients.

The combination of propofol and remifentanil is the most common in TIVA because of its fast pharmacokinetics and short half-life. However, the disadvantage of remifentanil is the lack of residual analgesic effect after termination of continuous infusion. As postoperative nasal packing can still bring postoperative pain, patients with severe discomfort caused by pain will have unexpected conditions such as surgical incision cracking and bleeding, which will affect the effect of operation and rehabilitation. Afentanil is another opioid drug with short effect and strong analgesic effect. Previous studies have shown that remifentanil-based TIVA has slightly higher postoperative pain and early use of analgesics than TIVA in discectomy. Because the effect of TIVA using Afentanil or remifentanil on postoperative pain in functional nasal endoscopic surgery is not clear, this study intends to observe the effect of TIVA on postoperative pain in patients undergoing functional nasal endoscopic surgery under general anesthesia, so as to optimize the clinical anesthetic scheme of this kind of minimally invasive surgery and provide clinical reference.

DETAILED DESCRIPTION:
This study intends to observe the effect of TIVA using afentanil or remifentanil on postoperative pain in patients undergoing functional nasal endoscopic surgery under general anesthesia.

Main indicators:

VAS score at 30 min after operation.

Secondary indicators:

VAS score of 60 min after operation. VAS score of 24h after operation. Number of cases of postoperative use of analgesics . Number of cases of postoperative adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* ASA Ⅰ-Ⅲ
* patients undergoing functional endoscopic sinus surgery under general anesthesia.

Exclusion Criteria:

* Significant hypertension (diastolic blood pressure > 100mmHg) or hypotension (systolic . blood pressure < 100mmHg).
* severe mental, cardiovascular, kidney or liver disease.
* previous history of alcohol or drug abuse.
* long-term use of painkillers before operation.
* contraindications for any drugs used in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
VAS score | Postoperative 30minutes
  the digital rating scale (VAS) uses a number between 0 and 10 to indicate that there is no pain; a score of 1-3 means that a slight pain can be tolerated; a score of 4-6 indicates that it is bearable if it does not affect sleep; a score of 7-10 indicates that it is becoming more and more painful and unbearable, affecting appetite and sleep

CONTACTS AND LOCATIONS:
Overall Officials: Yan Jia, Principal Investigator — The First Affiliated Hospital of the Air Force Medical Universtiy
Locations (1):
- YANLI, XIan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doganay G, Ekmekci P, Kazbek BK, Yilmaz H, Erkan G, Tuzuner F. Effects of alfentanil or fentanyl added to propofol for sedation in colonoscopy on cognitive functions: Randomized controlled trial. Turk J Gastroenterol. 2017 Nov;28(6):453-459. doi: 10.5152/tjg.2017.16489. Epub 2017 Sep 19. PMID 28928100
- See also: Doğanay G, Ekmekçi P, Kazbek BK, et al. Effects of alfentanil or fentanyl added to propofol for sedation in colonoscopy on cognitive functions: Randomized controlled trial. Turk J Gastroenterol. 2017 ,28(6):453-459. — https://pubmed.ncbi.nlm.nih.gov/28928100/